CLINICAL TRIAL: NCT03651388
Title: Research Into the Molecular Bases of a New Phenotype Combining Premature White Hair, Polycystic Kidney Disease, Aortic Dilation/Dissection and Lymphopenia
Acronym: BCL-2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER-FAIVRE AOI 2010
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: New Phenotype (Combining Premature White Hair, Polycystic Kidney Disease, Aortic Dilation/Dissection and Lymphopenia)
MeSH Terms: conditions — Polycystic Kidney Diseases; Lymphopenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patient with a new phenotype combining premature white hair, renal polycystosis, aortic dilation/dissection and lymphopenia
- Related parties of the 1st degree: 1st degree related family of Group A patient

SUMMARY:
This study involves a single family, including 1 patient, father, mother and sister. The patient presented with a new phenotype associating premature white hair, renal polycystosis, aortic dilation/dissection and lymphopenia. Samples were taken in order to identify the origin of the symptomatology highlighted in the index case.

In addition, it was observed that mice invalidated for bcl-2, normal at birth and indistinguishable from control mice, showed, after one week, a phenotype similar to that observed in this patient.

The overlap between the patient's main clinical signs (lymphopenia, white hair and polycystic renal disease) and the manifestations presented by the invalidated murine model for BCL2 suggests that its phenotype may be secondary to a Bcl-2 expression defect.

ELIGIBILITY:
This study involves a single family, including 1 patient, father, mother and sister.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patient
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Whole genome sequencing of BCL2 | Through study completion, an average of 2 years.
Bcl-2-regulating miRNA sequencing | Through study completion, an average of 2 years.
Study of the methylation of the BCL2 promoter | Through study completion, an average of 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France